CLINICAL TRIAL: NCT06536829
Title: Effects of Myofacial Release Technique With and Without Sciatic Nerve Slider Technique on Pain Range of Motion and Functional Disability Among Cricket Players With Sciatica.
Brief Title: Effects of Myofacial Release Technique and Sciatic Nerve Slider Technique in Sciatica
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR&AHS/23/0470
Record Dates: First submitted 2024-07-31; First posted 2024-08-05 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-07

CONDITIONS: Sciatic Neuropathy; Sciatica; Range of Motion
Keywords: Myofacial release tehnique (MFR), cricketer
MeSH Terms: conditions — Sciatic Neuropathy; Sciatica

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial.
Who Masked: Outcomes Assessor
Masking Description: single
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MYOFACIAL RELEASE TECHNIQUE, SCIATIC NERVE SLIDER TECHNIQUE (Experimental): Group A (18) and Group B(18). Both groups will be given a patient evaluation sheet. Group A will receive myofacial release technique and sciatic nerve slider technique with routine physiotherapy. simple myoficial release technique by applying gentle sustained pressure to the myoficial layer for 30-50 seconds. The myofacial release technique will apply on lumber region and calf musle. Group A will receive both techniques
  Interventions: Other: Myofacial release technique and sciatic nerve slider technique; Other: Myofacial release technique
- MYOFACIAL RELEASE TECHNIQUE (Experimental): Group B will receive just myofacial release technique and routine physiotherapy. Pain, range of motion and functional disability will be measured before session, immediate effect after first session, then after 06 weeks (18 session) and after weeks 12 (18 session) (3 sessions a week with 7-10 repetitions). with simple myoficial release technique by applying gentle sustained pressure to the myoficial layer for 30-50 seconds. The myofacial release technique will apply on lumber region and calf musle. Group B will receive myofacial release techniqe and routine physiotherapy.
  Interventions: Other: Myofacial release technique and sciatic nerve slider technique; Other: Myofacial release technique

INTERVENTIONS:
Other: Myofacial release technique and sciatic nerve slider technique — Myofacial release technique, sciatic nerve slider technique 0 week,6 week 12 weeks
  Other Names: routine physiotherpy
Other: Myofacial release technique — 0week,6 week, 12 weeks
  Other Names: Routine physiotherapy

SUMMARY:
Sciatica is not a medical condition itself, but is a symptom of whatever condition is affecting your sciatic nerve. Pain in the lower back, hip and legs is the most common symptom. However, tingling, numbness and weakness are also symptoms of a damaged sciatic nerve. Physical therapy is a popular and effective way of treating the pain from sciatica. Myofascial release (MFR) is another useful option for sciatica due to the fact that it focuses the connective tissues of the body, including muscles and the fibrous tissues, often called fascia, encircling the joints.This study will be conducted to compare the Effects of myofacial release technique with and without sciatic nerve slider technique on Pain, Range of Motion and Functional Disability among cricket players with Sciatica. This study will be conducted because, no such evidence found in literature to find out the effects of myofacial release technique with sciatic nerve slider technique for sciatica. Myofacial release technique and sciatic nerve slider technique are useful, because these can reduce patients number of visits for the treatment and are easy to use, feasible and cost effective. The sciatic nerve is the largest nerve in the human body. It is formed at the point where five nerves from the lower back all come together, and stretches all the way from the hips to the bottoms of the feet. When this important nerve becomes compressed, inflamed or irritated, it causes the pain in the lower back and legs known as sciatica. A physical therapist uses a number of proven methods to help relieve sciatic pain. One of the most commonly employed methods is known as myofascial release therapy. Myofascial release is a method that a physical therapist can use to treat many sources of pain that are caused by damage to the nervous system. It involves the therapist using hands-on, manual techniques to release areas of tension and pain in the body. Here are three reasons that myofascial release is an effective tool for treating sciatica.

DETAILED DESCRIPTION:
Physical therapy is a popular and effective way of treating the pain from sciatica. Myofascial release (MFR) is another useful option for sciatica due to the fact that it focuses the connective tissues of the body, including muscles and the fibrous tissues, often called fascia, encircling the joints.This study will be conducted to compare the Effects of myofacial release technique with and without sciatic nerve slider technique on Pain, Range of Motion and Functional Disability among cricket players with Sciatica. This study will be conducted because, no such evidence found in literature to find out the effects of myofacial release technique with sciatic nerve slider technique for sciatica. Myofacial release technique and sciatic nerve slider technique are useful, because these can reduce patients number of visits for the treatment and are easy to use, feasible and cost effective. The sciatic nerve is the largest nerve in the human body. It is formed at the point where five nerves from the lower back all come together, and stretches all the way from the hips to the bottoms of the feet. When this important nerve becomes compressed, inflamed or irritated, it causes the pain in the lower back and legs known as sciatica. A physical therapist uses a number of proven methods to help relieve sciatic pain. One of the most commonly employed methods is known as myofascial release therapy. Myofascial release is a method that a physical therapist can use to treat many sources of pain that are caused by damage to the nervous system. It involves the therapist using hands-on, manual techniques to release areas of tension and pain in the body. Here are three reasons that myofascial release is an effective tool for treating sciatica.

ELIGIBILITY:
Inclusion Criteria:

* Age group between 18-35 yrs.
* Male cricketers
* Pre diagnosed Patients suffering from sciatica referred from Orthopedic.
* History of low back pain atleast 03 months before enrollement.
* Pain while examing when straight leg test (SLR) is performed.
* Patients who are willing to particiapate in the study

Exclusion Criteria:

* History of any systemic disease
* History of trauma
* History of previous fracture in lower limb.
* History of prior Surgery
* Corticosteroid injection for lumber radiculopathy within previous 03 momths;
* Any known malignancy /neoplasma involved side.
* Diagnosed/known psychiatric illness.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — MALE
Enrollment: 36 (Estimated)
Dates: Start 2024-06-26 (Actual); Primary Completion 2024-09-26 (Estimated); Study Completion 2024-09-26 (Estimated)

PRIMARY OUTCOMES:
range of motion | 0 6 WEEKS 12 WEEKS
  will be measured Goniometer
Functional disability | 0 6 WEEKS 12 WEEKS
  will be measured LEFS

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Mohsin Raza, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Sports Board, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Geuna S. The sciatic nerve injury model in pre-clinical research. J Neurosci Methods. 2015 Mar 30;243:39-46. doi: 10.1016/j.jneumeth.2015.01.021. Epub 2015 Jan 25. PMID 25629799
- [Background] Mendez-Sanchez R, Alburquerque-Sendin F, Fernandez-de-las-Penas C, Barbero-Iglesias FJ, Sanchez-Sanchez C, Calvo-Arenillas JI, Huijbregts P. Immediate effects of adding a sciatic nerve slider technique on lumbar and lower quadrant mobility in soccer players: a pilot study. J Altern Complement Med. 2010 Jun;16(6):669-75. doi: 10.1089/acm.2009.0403. PMID 20569035
- [Background] Ahmad Siraj S, Dadgal R. Physiotherapy for Piriformis Syndrome Using Sciatic Nerve Mobilization and Piriformis Release. Cureus. 2022 Dec 26;14(12):e32952. doi: 10.7759/cureus.32952. eCollection 2022 Dec. PMID 36712711
- [Background] Ozsoy G, Ilcin N, Ozsoy I, Gurpinar B, Buyukturan O, Buyukturan B, Kararti C, Sas S. The Effects Of Myofascial Release Technique Combined With Core Stabilization Exercise In Elderly With Non-Specific Low Back Pain: A Randomized Controlled, Single-Blind Study. Clin Interv Aging. 2019 Oct 9;14:1729-1740. doi: 10.2147/CIA.S223905. eCollection 2019. PMID 31631992